CLINICAL TRIAL: NCT07160452
Title: Effect of Levocarnitine Injections on Reducing Erythropoietin-Stimulating Agent Requirements in Hemodialysis Patients With Renal Anemia
Brief Title: Levocarnitine for Reducing ESA Requirements in Hemodialysis Patients With Renal Anemia
Acronym: L-CAR-ESA
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shaikh Zayed Hospital, Lahore (Other)
Responsible Party: Principal Investigator, Hanzla Arshad, Doctor, Shaikh Zayed Hospital, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TERC/SC/INT/2025/455
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Anemia; Kidney Failure; End-Stage Renal Disease; Renal Dialysis
Keywords: Levocarnitine; L-carnitine; Erythropoiesis-Stimulating Agents; Erythropoietin Responsiveness Index; Hematocrit
MeSH Terms: conditions — Anemia; Renal Insufficiency; Kidney Failure, Chronic | interventions — Carnitine

STUDY DESIGN:
Intervention Model Description: Single-center, two-arm, open-label, randomized controlled trial with 1:1 allocation by simple randomization (lottery). Adults on maintenance hemodialysis with renal anemia are assigned to levocarnitine 1,000 mg IV three times weekly after dialysis plus usual ESA care versus usual ESA care without levocarnitine. Follow-up 6 months; monthly assessments of Hb, Hct, ESA dose, and ERI.
Masking Description: Open-label; no parties masked. Primary outcomes (ESA dose, ERI, Hb/Hct) are obtained from routine records.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levocarnitine + Usual ESA Care (Experimental): Adults on maintenance hemodialysis with renal anemia receive levocarnitine 1,000 mg IV immediately after each dialysis session, three times per week for 6 months, in addition to standard anemia management with erythropoiesis-stimulating agents (ESA) per unit protocol. Monthly assessments of hemoglobin, hematocrit, ESA dose, and erythropoietin responsiveness index (ERI).
  Interventions: Drug: Levocarnitine Injection; Other: Usual ESA-Based Anemia Care
- Usual ESA Care (No Levocarnitine) (Active Comparator): Standard anemia management with ESA per unit protocol without levocarnitine. Monthly assessments of hemoglobin, hematocrit, ESA dose, and ERI over 6 months.
  Interventions: Other: Usual ESA-Based Anemia Care

INTERVENTIONS:
Drug: Levocarnitine Injection — 1,000 mg levocarnitine IV (slow IV push or infusion per unit policy) post-hemodialysis, three times weekly for 6 months (~72 doses). Administered in the dialysis unit in addition to usual ESA-based anemia care.
  Other Names: L-carnitine; Levocarnitine; Carnitine
  Arms: Levocarnitine + Usual ESA Care
Other: Usual ESA-Based Anemia Care — Standard-of-care anemia management using recombinant human erythropoietin (ESA) per unit protocol. Typical initial dosing: 50-100 U/kg/week if Hb <10 g/dL (in 2-3 doses/week); 50 U/kg/week if Hb 10-11 g/dL; 25-50 U/kg/week as maintenance if Hb 11-12 g/dL. ESA dose adjusted monthly using ERI and Hb/Hct targets (generally Hb 10-12 g/dL).

SUMMARY:
Renal anemia is common in people receiving long-term hemodialysis and is usually treated with erythropoiesis-stimulating agents (ESAs). Some patients respond poorly and require high ESA doses, which increases treatment burden, cost, and potential side effects. Carnitine deficiency is frequent in hemodialysis because carnitine is lost during dialysis and its synthesis is reduced. Levocarnitine may improve red blood cell function and reduce the dose of ESA needed to maintain hemoglobin.

This single-center, randomized controlled trial will test whether adding intravenous levocarnitine to standard care reduces ESA requirements in adults on maintenance hemodialysis who have renal anemia. Ninety-four participants (age 20-60 years) on thrice-weekly hemodialysis for ≥6 months and with hemoglobin <10 g/dL will be randomly assigned (1:1) to:

Intervention: Levocarnitine 1,000 mg IV three times per week, administered after each dialysis session, plus usual anemia care including ESA per unit protocol.

Control: Usual anemia care including ESA per unit protocol without levocarnitine.

Participants will be followed for 6 months. Hemoglobin, hematocrit, ESA dose, and the erythropoietin responsiveness index (ERI = monthly ESA dose ÷ [dry weight × average hemoglobin]) will be recorded monthly.

The primary outcome is the ESA dose (units/week) at month 6. Secondary outcomes include ERI and monthly changes in hemoglobin and hematocrit, along with routine safety monitoring. If levocarnitine lowers ESA needs, the findings may offer a cost-effective strategy to optimize anemia management in hemodialysis patients.

DETAILED DESCRIPTION:
Background and Rationale. Carnitine supports erythrocyte membrane stability and energy metabolism. In maintenance hemodialysis, endogenous carnitine synthesis is reduced and dialytic losses occur, potentially contributing to ESA hyporesponsiveness. Small trials suggest that levocarnitine may reduce ESA dose requirements while maintaining target hemoglobin. Robust, region-specific evidence is limited.

Study Overview. This is a single-center, two-arm, randomized (1:1), open-label, parallel-group trial conducted at the Department of Nephrology, Shaikh Zayed Hospital, Lahore. Adults on thrice-weekly maintenance hemodialysis are randomized to: (A) adjunct levocarnitine 1,000 mg IV after each dialysis session, or (B) standard care without levocarnitine. ESA therapy is provided to all participants according to institutional practice, with dose adjustments based on routine hemoglobin monitoring. Study follow-up is 6 months, with monthly assessments of laboratory indices and ESA use. Full eligibility criteria, outcome measures (including the definition of the erythropoietin responsiveness index), intervention details, and visit schedule are specified in the corresponding PRS modules.

Statistical Considerations. The trial is powered (80% at α=0.05) to detect a between-group difference in ESA use at 6 months based on prior data; the planned sample size is 94 participants (47 per group). Analyses will follow the intention-to-treat principle, with supportive per-protocol analyses. Continuous outcomes will be summarized as mean±SD or median [IQR], and compared using appropriate two-sample methods. Prespecified subgroup and sensitivity analyses may adjust for baseline factors such as age, sex, BMI, and comorbidity status.

Safety and Monitoring. Adverse events and intercurrent illnesses are captured at each visit and via clinical record review. Any clinically significant events will be reported per institutional procedures. Data will be recorded on standardized case-report forms and managed to protect participant confidentiality.

Significance. Demonstrating reduced ESA requirements with levocarnitine while maintaining target hemoglobin could improve patient care and lower treatment costs in resource-constrained dialysis programs.

ELIGIBILITY:
Inclusion Criteria:

1. Both male and female patients
2. Patients aged 20-60 years.
3. Patients undergoing maintenance hemodialysis three times a week for at least six months
4. Patients having renal anemia

Exclusion Criteria:

1. Patients currently using any carnitine preparation as a supplement (to avoid confounding effects from additional carnitine intake).
2. Patients on immunosuppressive drugs, steroids, or antibiotics (to avoid the influence of these medications on anemia and carnitine metabolism).
3. Patients who have previously received levocarnitine in either oral or injected form (to eliminate any prior influence of levocarnitine on study outcomes).
4. Patients with a history of blood transfusion within the past 6 months (to exclude the immediate impact of transfusions on hemoglobin levels and anemia management).
5. Patients with acute inflammation (to prevent interference with study parameters as inflammation can affect anemia status).
6. Patients with communication difficulties due to dementia or other factors (to ensure accurate symptom reporting and study adherence).

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Weekly ESA dose at Month 6 (units/week) | Month 6 (plus or minus 2 weeks) after randomization
  Total weekly dose of erythropoiesis-stimulating agent (ESA; recombinant human erythropoietin or biosimilar) abstracted from the dialysis unit medication administration record. Recorded as the sum of ESA units administered in the 7-day period closest to the Month-6 visit. Lower values indicate an ESA-sparing effect.

SECONDARY OUTCOMES:
Change in weekly ESA dose from Baseline to Month 6 (units/week) | Baseline and Month 6 (±2 weeks)
  Difference = (Month-6 weekly ESA dose) - (Baseline weekly ESA dose), from medication records. Negative values indicate dose reduction.

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the published results will be available to qualified researchers upon reasonable request after publication of the primary manuscript.
Supporting Information: SAP, ICF
Time Frame: From 12 months after publication for up to 5 years.
Access Criteria: Requests with a methodologically sound proposal, protocol, and analysis plan should be directed to the Principal Investigator. Data access will require IRB/ethics approval (if applicable) and a data use agreement.

REFERENCES:
- [Background] Morgans HA, Chadha V, Warady BA. The role of carnitine in maintenance dialysis therapy. Pediatr Nephrol. 2021 Aug;36(8):2545-2551. doi: 10.1007/s00467-021-05101-z. Epub 2021 Jun 18. PMID 34143302
- [Background] Kadiroglu AK, Yilmaz ME, Sit D, Kara IH, Isikoglu B. The evaluation of postdialysis L-carnitine administration and its effect on weekly requiring doses of rHuEPO in hemodialysis patients. Ren Fail. 2005;27(4):367-72. PMID 16060121
- [Background] Maruyama T, Higuchi T, Yamazaki T, Okawa E, Ando H, Oikawa O, Inoshita A, Okada K, Abe M. Levocarnitine Injections Decrease the Need for Erythropoiesis-Stimulating Agents in Hemodialysis Patients with Renal Anemia. Cardiorenal Med. 2017 Jun;7(3):188-197. doi: 10.1159/000462983. Epub 2017 Apr 20. PMID 28736559